CLINICAL TRIAL: NCT06022081
Title: Comparative Evaluation of Novice-Performed Lung Ultrasound vs. Chest X-Ray for Pneumothorax Detection Post-Chest Tube Removal in Cardiac Surgery and Trauma Patients
Brief Title: Lung Ultrasound Versus Chest Radiography for Detection of Pneumothorax
Acronym: LUSvsCXR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Jacobo Moreno Garijo, Staff Anesthesiologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5854
Record Dates: First submitted 2023-08-16; First posted 2023-09-01 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pneumothorax
Keywords: Pneumothorax; Lung Ultrasound; Chest X-Ray; Trauma patients; Cardiac Surgery; Chest Drain Removal
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Intervention Model Description: Single-group study where the focus is on evaluating the diagnostic accuracy of both CXR and LUS for PNX detection post-tube removal in cardiac surgery and trauma patients. The study aims to compare the results of both modalities within the same group of participants to assess their performance in detecting PNX.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic modalities comparison (Other): All participants belong to a single arm. A chest X-ray (CXR) and lung ultrasound (LUS) in a predetermined order (CXR followed by LUS), will be performed sequentially for pneumothorax (PNX) detection after chest/mediastinal tube removal. There is no control group or randomization.
  Interventions: Diagnostic Test: Lung ultrasound to detect pneumothorax.

INTERVENTIONS:
Diagnostic Test: Lung ultrasound to detect pneumothorax. — Within a maximum of two hours after chest tube removal, the sonographic exam will be performed with an ultrasound device to assess residual PNX using a portable ultrasound device. The examination will require patients to lie face upward and will be performed at three different sites on both sides of the patient's chest. Each chest site will be imaged for approximately 10-20 seconds, allowing a complete examination of each side in approximately 30-60 seconds. The total study time for the LUS exam is approximately 2 minutes. The results of this assessment will be compared to the standard chest x-ray performed by a radiologist who is unaware of the study.

SUMMARY:
Sunnybrook Health Sciences Center annually provides assistance to approximately 600 cardiac surgeries and 1500 trauma patients, many of whom require chest tubes to prevent blood and fluids from accumulating in the pleural cavities surrounding the heart. During the removal of chest tubes, there is a risk of air leaking into these cavities, leading to pneumothorax, a critical condition occurring in approximately 5-26% of cases, associated with increased complications and mortality.

Currently, the diagnosis of pneumothorax is primarily based on chest X-rays (CXR), despite their limitations and low reliability. As an alternative method, lung ultrasound (LUS) offers several advantages: it is safer, less expensive, and less painful for patients compared to CXR. However, there is a lack of comparative data on the accuracy and interrater reliability of these two diagnostic approaches after chest tube removal.

This study aims to evaluate the accuracy of lung ultrasound performed by medical trainees in diagnosing pneumothorax in cardiac and trauma patients. By comparing LUS to CXR, the investigators seek to determine if LUS provides a more reliable and precise diagnosis. This study has the potential to enhance patient care by establishing a more effective and accessible method for diagnosing pneumothorax post-chest tube removal.

DETAILED DESCRIPTION:
Diagnosing and promptly treating pneumothorax (PNX) is critical, as it is associated with increased morbidity, mortality, and hospital stay for patients. Following cardiac surgery, timely identification of PNX is particularly vital due to patients' reduced cardiopulmonary reserve, which can rapidly lead to life-threatening situations. While computed tomography (CT) is highly accurate in diagnosing PNX, its routine use for screening is impractical due to high radiation exposure, cost, and limited availability. Currently, the standard method for PNX detection is chest X-ray (CXR), but its reliability is suboptimal, resulting in potential misdiagnoses and delays in patient care.

An alternate method for detecting PNX is using lung ultrasound (LUS). LUS is safe, portable compared to CXR, has the potential for faster results and higher accuracy relative to CXR. LUS can also be carried out by appropriate trained nurses and medical trainees, instead of requiring an expert radiographer. This prospective, single-center, observational, cross-sectional, cohort, feasibility pilot trial assesses trainee-performed bedside lung ultrasound (LUS) for detecting PNX and testing feasibility for a multicenter observational prospective study.

The investigators will also compare PNX detection using LUS by novices compared to experts, interrater reliability and the time required from chest/mediastinal tube removal to diagnostic report for LUS. All participants will undergo assessment for PNX using both LUS and CXR completed independently (by study-trained critical care nurse/surgical trainee or an expert radiologist, respectively) and results will be compared between the two modalities.

The successful implementation of LUS could lead to streamlined patient care and improved outcomes for cardiac surgery and trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Cardiac and trauma patients who have had a chest/mediastinal tube removed within the past two hours in the CVICU, trauma bay, or ward.

Exclusion Criteria:

* Patients who had a PNX prior to mediastinal chest tube removal that required intervention.
* Patients on mechanical ventilation.
* Patients with subcutaneous emphysema due to impaired pleural line visualization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 12 months (full pilot trial)
  The total number of participants recruited during the pilot trial. Target: 60 participants.
Adherence to LUS Scan Protocol | 12 months (full pilot trial)
  The proportion of participants who receive the LUS scans as per the trial protocol. This will be assessed by checking the frequency of LUS scans conducted for each participant against the planned frequency in the protocol. Measurement Tool: Frequency count of LUS scans against planned protocol scans.
Feasibility of Accurate LUS Data Collection for Comparison with Chest X-rays | 12 months (full pilot trial)
  Evaluate the feasibility of obtaining accurate LUS data suitable for comparison against Chest X-rays. The accuracy of LUS scans will be determined by the clarity and consistency of recorded data points. For the purpose of this study, 'accuracy' will be defined by a set of criteria based on sonographic signs of pneumothorax that include: absence of lung sliding, absence of B lines, presence of lung point, and absence of lung pulse. The primary outcome will be the proportion of LUS scans that meet this accuracy threshold. Measurement Tool: Qualitative assessment criteria tailored for this study. LUS scans will be evaluated based on clarity, consistency of recorded data points, and adherence to the sonographic signs of pneumothorax as listed above. The results from LUS will then be prepared for comparison against Chest X-ray findings in subsequent analyses.

SECONDARY OUTCOMES:
Compare novice-performed LUS with CXR reports performed by experienced radiologists. | 12 months (full pilot trial)
  The results of the assessments will be analyzed to determine the sensitivity, specificity, positive predictive value, and negative predictive value of pneumothorax detection by novices compared to experts.
Diagnostic accuracy of LUS vs CXR | 12 months (full pilot trial)
  Assess diagnostic accuracy and sensitivity of PNX detection by CXR and LUS (80% interrater reliability with the results when LUS is adjudicated by an expert for detecting PNX post-chest/mediastinal tube removal).
Diagnostic Sensitivity of CXR vs LUS | 12 months (full pilot trial)
  Assess diagnostic sensitivity of PNX detection by CXR and LUS (80% interrater reliability with the results when LUS is adjudicated by an expert for detecting PNX post-chest/mediastinal tube removal).
Interrater reliability | 12 months (full pilot trial)
  Assess the interrater reliability of novice and expert sonographers.
Time Required | 12 months (full pilot trial)
  Assess the time required from chest/mediastinal tube removal to diagnostic report for LUS vs CXR.

CONTACTS AND LOCATIONS:
Overall Officials: Jacobo Moreno Garijo, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Science Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon publication, no limit on time
Access Criteria: Contact study investigators

REFERENCES:
- [Background] Khan T, Chawla G, Daniel R, Swamy M, Dimitri WR. Is routine chest X-ray following mediastinal drain removal after cardiac surgery useful? Eur J Cardiothorac Surg. 2008 Sep;34(3):542-4. doi: 10.1016/j.ejcts.2008.05.002. Epub 2008 Jun 9. PMID 18539477
- [Background] Bell RL, Ovadia P, Abdullah F, Spector S, Rabinovici R. Chest tube removal: end-inspiration or end-expiration? J Trauma. 2001 Apr;50(4):674-7. doi: 10.1097/00005373-200104000-00013. PMID 11303163
- [Background] McCormick JT, O'Mara MS, Papasavas PK, Caushaj PF. The use of routine chest X-ray films after chest tube removal in postoperative cardiac patients. Ann Thorac Surg. 2002 Dec;74(6):2161-4. doi: 10.1016/s0003-4975(02)03982-6. PMID 12643411
- [Background] Pacharn P, Heller DN, Kammen BF, Bryce TJ, Reddy MV, Bailey RA, Brasch RC. Are chest radiographs routinely necessary following thoracostomy tube removal? Pediatr Radiol. 2002 Feb;32(2):138-42. doi: 10.1007/s00247-001-0591-5. Epub 2001 Nov 24. PMID 11819085
- [Background] Goodman MD, Huber NL, Johannigman JA, Pritts TA. Omission of routine chest x-ray after chest tube removal is safe in selected trauma patients. Am J Surg. 2010 Feb;199(2):199-203. doi: 10.1016/j.amjsurg.2009.03.011. PMID 20113700
- [Background] Eisenberg RL, Khabbaz KR. Are chest radiographs routinely indicated after chest tube removal following cardiac surgery? AJR Am J Roentgenol. 2011 Jul;197(1):122-4. doi: 10.2214/AJR.10.5856. PMID 21701019
- [Background] Diaz R, Patel KB, Almeida P, Shekar SP, Hernandez F, Mehta JP. Are Chest Radiographs Routinely Indicated After Chest Tubes Placed for Non-Surgical Reasons Are Removed? Cureus. 2020 Mar 20;12(3):e7339. doi: 10.7759/cureus.7339. PMID 32313780
- [Background] Tocino IM, Miller MH, Fairfax WR. Distribution of pneumothorax in the supine and semirecumbent critically ill adult. AJR Am J Roentgenol. 1985 May;144(5):901-5. doi: 10.2214/ajr.144.5.901. PMID 3872573
- [Background] Galbois A, Ait-Oufella H, Baudel JL, Kofman T, Bottero J, Viennot S, Rabate C, Jabbouri S, Bouzeman A, Guidet B, Offenstadt G, Maury E. Pleural ultrasound compared with chest radiographic detection of pneumothorax resolution after drainage. Chest. 2010 Sep;138(3):648-55. doi: 10.1378/chest.09-2224. Epub 2010 Apr 9. PMID 20382717
- [Background] Ball CG, Kirkpatrick AW, Feliciano DV. The occult pneumothorax: what have we learned? Can J Surg. 2009 Oct;52(5):E173-9. PMID 19865549